CLINICAL TRIAL: NCT02579993
Title: ABCB5 as a Prognostic Marker in Survival of Cultivated Limbal Stem Cell Transplantation Expanded in Vitro on Amniotic Membrane in Patients With Limbal Stem Cell Deficiency.
Brief Title: ABCB5 as a Prognostic Marker in Survival of Cultivated Limbal Stem Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminar results not favorable
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-051-2014
Record Dates: First submitted 2015-10-11; First posted 2015-10-20 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: Cornea; Limbal stem cell
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Transplantation (Experimental): Cultivated Limbal Stem Cell Transplantation
  Interventions: Procedure: Pannus and conjunctival dissection; Procedure: Human cultivated limbal stem cell transplantation

INTERVENTIONS:
Procedure: Pannus and conjunctival dissection — A complete conjunctival peritomy is performed and the fibrovascular pannus and conjunctiva invading the cornea is dissected from the cornea and limbus.
Procedure: Human cultivated limbal stem cell transplantation — The amniotic membrane graft cultured with the human limbal stem cell transplantation is placed in the limbic and corneal surface and fixed with fibrin glue. The amniotic membrane is placed with the stroma in contact with the graft and it is sutured.

SUMMARY:
In this study the prognostic value of ABCB5 in survival of the limbal stem cell transplantation expanded in vitro on amniotic membrane for corneal surface reconstruction in patients with limbal stem cell deficiency will be analyzed.

DETAILED DESCRIPTION:
There are several diseases that cause the cornea to lose its clarity and directly affects the vision of the individual, therefore, the use of limbal stem cells has been having increasing acceptance in the field of medical therapy. An open clinical study is running with patients with limbal stem cell deficiency, performing a limbal stem cell transplantation expanded in vitro on amniotic membrane and the value of ABCB5 as a prognostic factor in the survival of transplant will be determined. The corneal surface status will be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral limbal stem cell deficiency of any etiology.
2. Corneal impression cytology positive for goblet cells.
3. Ocular ultrasound results within normal parameters.
4. Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Active immunological diseases.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Objective clinical evaluation | 6 months
  A grading system from 0 to 4 using photographs taken with slit lamp, will be used to determine by two independent examiners the degree of corneal transparency and superficial vascularization.
Objective clinical evaluation | 12 months
  A grading system from 0 to 4 using photographs taken with slit lamp, will be used to determine by two independent examiners the degree of corneal transparency and superficial vascularization.

SECONDARY OUTCOMES:
Corneal cells morphology | 6 months
  Evaluation of the presence of epithelial, conjunctival or mixed cells with in vivo confocal microscopy and impression cytology
Corneal cells morphology | 12 months
  Evaluation of the presence of epithelial, conjunctival or mixed cells with in vivo confocal microscopy and impression cytology
Quality of life questionnaire | 6 months
  Modified National Eye Institute Visual Function Questionnaire 25 questionnaire
Quality of life questionnaire | 12 months
  Modified National Eye Institute Visual Function Questionnaire 25 questionnaire
Visual acuity | 6 months
  Visual acuity in the Logarithm of the Minimum Angle of Resolution scale
Visual acuity | 12 months
  Visual acuity in the Logarithm of the Minimum Angle of Resolution scale

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Garfias, MD, PhD, Study Director — Instituto de Oftalmologia Conde de Valenciana
Locations (1):
- Instituto de Oftalmologia Conde de Valenciana, Mexico City, Mexico

REFERENCES:
- [Derived] Serna-Ojeda JC, Garcia-Mejia M, Graue-Hernandez EO, Navas A, Garfias Y. Short-Term Results Analysis in the Allogenic Transplantation of Limbal Stem Cells Expanded on Amniotic Membrane in Patients with Bilateral Limbal Stem Cell Deficiency. J Ocul Pharmacol Ther. 2020 May;36(4):238-246. doi: 10.1089/jop.2019.0147. Epub 2020 Feb 20. PMID 32077779